CLINICAL TRIAL: NCT01220960
Title: A Mixed Methods Approach to Evaluating How Art Therapy Can Benefit Women Recently Diagnosed With Breast Cancer
Brief Title: Art Therapy Intervention for Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Sarkis Meterissian (Other)
Collaborators: The Cedars Cancer Institute (Unknown)
Responsible Party: Sponsor-Investigator, Dr. Sarkis Meterissian, Professor of Surgery and Oncology Clinic, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 10-049-PSY
Record Dates: First submitted 2010-10-09; First posted 2010-10-14 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: Breast Cancer
Keywords: art therapy; breast cancer; women; young women; older women; quality of life; meaning making; support group; art making; art symbols
MeSH Terms: conditions — Breast Neoplasms | interventions — Art Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Art Therapy intervention group (Experimental): For participants who will be part of the art therapy intervention, the art therapy group will be a closed group for eight women with breast cancer who are in treatment and recently have had surgery. The group will meet once a week for two hours over a period of 8 weeks, and will focus on exploring the expressive capabilities of art making in a supportive group. This group will be held in the conference room at the Cedars Breast Clinic. Each week will revolve around a theme that pertains to the experience of women living with breast cancer, and will be guided by the women's needs in the group. A broad range of art materials will be made available and various art techniques explored. No art experience is necessary. The intervention group will also need to fill out simple questionnaires before the art therapy groups starts and after the group finishes
  Interventions: Other: art therapy
- Control Group (No Intervention): The group not assigned to the intervention group will be asked to fill out questionnaires at two separate times (before and after the intervention group is run). The Control group will be offered the opportunity to join an open art therapy group upon completing the questionnaires.

INTERVENTIONS:
Other: art therapy — Art therapy sessions, 2 hours in duration, 1 session/week, 8 continuous weeks of sessions. Each group will be limited to eight women as space is limited.
  Arms: Art Therapy intervention group

SUMMARY:
As studies continue to debate the effects of quality of life on survival, increased attention is being focused on investigating complementary alternative therapies to boost overall total health in cancer patients . Art therapy is an interesting growing field, which has shown promise to positively influence quality of life in the pediatric and adult oncology population alike. As there is a paucity of well controlled complete studies in this field, the investigators propose to study the impact of art therapy sessions in women with breast cancer with quantitative and qualitative analysis of emotional health and physical symptoms.

The results of the investigators study will have widespread applicability to oncology programs that wish to offer/implement such sessions to their palliative and non-palliative outpatients in an effort to address the important concept of whole person care.

ELIGIBILITY:
Inclusion Criteria:

1. Any woman 18-years or older
2. Stage I to III breast cancer (first time diagnosis)
3. Minimum of 6 weeks Post Operative status

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2010-08; Primary Completion 2012-12 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Quality of Life (emotional distress, physical symptoms,self-efficacy and well-being) | 8 weeks
  To investigate whether the implementation of an 8 week art therapy course in post-operative outpatient breast cancer patients can alleviate/improve
  1. Emotional distress as assessed by the Hospital Depression and Anxiety Scale (HADS) (please see below for details)
  2. Physical symptoms as assessed by the Edmonton Symptom Assessment Scale (ESAS)
  3. Meaning making as assessed by The Generalized Self-Efficacy Scale (GSES) and the Functional Assessment of Chronic Illness Therapy-Spiritual Well-Being Scale (FACIT-Sp-12).

SECONDARY OUTCOMES:
Ability to find and create meaning after the psychosocial impact of a breast cancer diagnosis | 8 weeks
  To investigate qualitatively how group art therapy can address the psychosocial impacts of breast cancer, including the challenges of finding and creating meaning following a recent diagnosis of breast cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine L Laux, MA Art Therapy, Principal Investigator — Cedars CanSupport; Virginia Lee, PhD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Sharon Wexler, PhD, Principal Investigator — Cedars CanSupport; Monisha Sudarshan, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Sarkis Meterissian, PhD, Study Director — MUHC Cedars Breast Centre
Locations (1):
- Cedars Breast Centre\ Royal Victoria Hospital, Montreal, Quebec, Canada